CLINICAL TRIAL: NCT00481013
Title: Prospective Controlled Trial of Valproic Acid in Ambulant Adults With Spinal Muscular Atrophy (VALIANTSMA) Study
Brief Title: Valproic Acid in Ambulant Adults With Spinal Muscular Atrophy
Acronym: VALIANTSMA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Families of Spinal Muscular Atrophy (Other); Abbott (Industry)
Responsible Party: Principal Investigator, Kathryn Swoboda, Associate Professor, Neurology and Pediatrics, University of Utah
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2006H0249
Record Dates: First submitted 2007-05-30; First posted 2007-06-01 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Spinal Muscular Atrophy
Keywords: Spinal Muscular Atrophy; Adult
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — Valproic Acid; Carnitine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1a (Placebo Comparator): For six months, half of patients are randomized into placebo . After 6 months, all patients are on treatment.
  Interventions: Drug: Placebo
- 1b (Active Comparator): Cohort 1b patients are randomized onto treatment. After 6 months, all patients are on drug.
  Interventions: Drug: Valproic Acid (VPA)

INTERVENTIONS:
Drug: Valproic Acid (VPA) — Drug: Valproic Acid and Levocarnitine; capsules
  Other Names: Depakote; Carnitor
  Arms: 1b
Drug: Placebo — For six months, pts are randomized into placebo or treatment. After 6 months, all pts are on treatment
  Arms: 1a

SUMMARY:
The primary objective of this proposal is to determine whether oral VPA is effective in treating SMA in adult patients.

DETAILED DESCRIPTION:
Participation in this study entails six visits and seven to eight blood draws over 13 months. Each visit entails a stay of two days and one night at the General Clinical Research Center (GCRC).

Subjects who live within driving distance will be allowed to participate in the study without an overnight stay through two consecutive outpatient visits. All subjects will be evaluated at two screening visits 2-4 weeks apart to determine eligibility for participation. Eligible subjects will be randomized to receive VPA or placebo for the first six months. At the six-month visit, patients will be evaluated and crossed over to the other regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory adults with SMA 3 ages 18-60. The diagnosis of SMA must be documented by the homozygous deletion of both SMN1 genes on standard genetic tests for the disorder. Patients must be able to walk thirty feet without assistance (i.e. no canes, walkers).
2. Interest in participating and the ability to meet the study requirements.
3. Women of child bearing age are required to be on birth control or abstain while participating in the study.

Exclusion Criteria:

1. Non-ambulatory type 3 adults and all type 2 adults.
2. Patients with co-morbid conditions that preclude travel, testing or study medications.
3. Patients who have participated in a treatment trial for SMA in the 3 months prior to this trial, or plan on enrolling in any other treatment trial during the duration of this trial.
4. Patients who are, in the investigator's opinion, mentally or legally incapacitated from providing informed consent for the study, or are otherwise unable to meet study requirements or cooperate reliably with study procedures, especially strength testing.
5. Patients with a need for non-invasive ventilatory support (e.g. BiPAP) for > 12 hours/day
6. Transaminases, amylase or lipase > 3.0 x normal values, WBC < 3.0 or neutropenia < 1.0, platelet count < 100 K, or hematocrit < 30 persisting over a 30 day period
7. Use of medications or supplements which interfere with VPA metabolism and increase the potential risks of the medications, or are hypothesized to have a beneficial effect in SMA animal models or human neuromuscular disorders within 3 months of study enrollment. These agents include riluzole, creatine, butyrate derivatives, growth hormone, anabolic steroids, daily albuterol use, anticonvulsants, or other HDAC inhibitors.
8. Women who are pregnant or who intend to become pregnant while participating in the research study or who are breastfeeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2007-07; Primary Completion 2009-12 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
The primary outcome for the study is change in muscle strength from baseline to six months in muscle strength as assessed by MVICT using a fixed testing system. | 13 months

SECONDARY OUTCOMES:
Change in SMAFRS | 13 months
Change in strength assessed by hand-held dynamometer | 13 months
Change in MUNE and CMAP | 13 months
SMN2 copy number | 13 months
Change in PFTs, including forced vital capacity (FVC) and negative inspiratory force (NIF) | 13 months
Change in lean body mass through DEXA scanning | 13 months
Change in distance walked in 6 minutes | 13 months
Change in time to climb four standard stairs | 13 months
Change in health-related QOL assessed through the modified sickness impact profile (SIP) | 13 months

CONTACTS AND LOCATIONS:
Overall Officials: John T Kissel, Principal Investigator — Ohio State University; Sandra P Reyna, M.D., Study Director — Families of Spinal Muscular Atrophy; Kathryn J Swoboda, M.D., Principal Investigator — University of Utah
Locations (1):
- Ohio State University Medical Center, Dept. of Neurology, Columbus, Ohio, United States